CLINICAL TRIAL: NCT04598360
Title: A Lipidomics Study: Release of Epoxyeicosatrienoic Acids From Erythrocytes During the Use of Extracorporeal Procedures (Heart-lung Machine)
Brief Title: Release of Epoxyeicosatrienoic Acids From Erythrocytes During the Use of Extracorporeal Procedures (Heart-lung Machine)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, Benjamin Gollasch, Benjamin Gollasch, Charite University, Berlin, Germany
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: EA2/113/08
Record Dates: First submitted 2020-10-16; First posted 2020-10-22 (Actual); Last update posted 2022-03-22 (Actual); Status verified 2022-03

CONDITIONS: Coronary Arteriosclerosis; Valve Heart Disease
Keywords: Fatty Acid Metabolism; Erythrocytes; Lipidomics; Heart-Lung-Machine
MeSH Terms: conditions — Coronary Artery Disease; Heart Valve Diseases | interventions — Heart-Lung Machine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental: Erythrocyte Fatty-Acid Status (Experimental): Erythrocyte Fatty-Acid Status Profiling of cardiac surgery patients are studied before and during heart-lung-machine procedure using LC-MS / MS
  Interventions: Procedure: Heart-Lung-Machine

INTERVENTIONS:
Procedure: Heart-Lung-Machine — blood sample before and during a single Heart-Lung-Machine procedure

SUMMARY:
Hypotension with potentially serious consequences for organ perfusion is a common complication in extracorporeal procedures such as heart-lung-machine. The exact reasons for this are still insufficiently clarified. Probably periinterventional vasorelaxant released substances play a crucial role in these procedures. These substances could be due to contact of blood cells with the Membrane in the HLM arise. In this project the hypothesis will be checked, if EETs / DHETs are released by Erythrocytes during this extracorporeal procedure and thus act as potential candidate products for the result of hypotonic phases during usage of heart-lung-machine.

We will determine differences in RBC fatty acids profiling in patients before and after heart-lung-machine intervention. RBC fatty acids profiling will be achieved by using targeted HPLC-MS mass spectrometry.

It is believed that during HLM there is an increase in EETs / DHETs in the serum and in the erythrocytes. It is believed that shear forces play an important role in the release of erythrocyte EETs / DHETs.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are undergoing an operation with the aid of the heart-lung machine for cardiac surgery
* Age over 18 years
* Ability to consent
* There is a written consent of the study participant

Exclusion Criteria:

•none

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2020-11-01 (Actual); Primary Completion 2021-09-01 (Actual); Study Completion 2022-01-01 (Actual)

PRIMARY OUTCOMES:
Coefficient of variation of relative quantities of erythrocyte fatty-acid parameters related to its dynamic during HLM, using LC-MS / MS. | 4-5months
  EETs / DHETs will be analyzed in the erythrocytes and serum of the recovered blood samples.
  The determination will made in cooperation with a Berliner Biotech company. This involves liquid chromatography with MS coupling (LC-MS / MS) used. The data analysis is carried out by means of suitable statistical methods to perform erythrocyte fatty-acid status profiling.

CONTACTS AND LOCATIONS:
Locations (1):
- Charité University Experimental & Clinical Research Center, Berlin, Germany

IPD SHARING:
Plan to Share IPD: Undecided